CLINICAL TRIAL: NCT01228487
Title: Biomechanical Factors of Secondary Osteoarthritis: Oxidative and Nitrosative Stress as Predictive Factors of Joint Destruction
Brief Title: Influence of Oxidative Dysbalance on Secondary Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Prof. Dr. med. R. Krauspe, Head of Orthopaedic Department, Heinrich-Heine University, Duesseldorf
Other Study IDs: ORTH-OA-1
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Osteoarthritis
Keywords: Oxidative Dysbalance; Oxidative Stress; Biomarker
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arthroscopical obtained wash- out preparations of synovial space Synovial biopsies Blood serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute knee pain: Patients with a history of knee pain < 6 months. The radiologic and arthroscopic OA stadium is less or equal II°. n=20.
- Chronic knee pain: Clinical manifestation of knee joint OA, radiological and arthroscopic III° or more. n=20
- Control group: Patients coming for post- primary repair of the cruciate ligament, having no inflammation and no sign of OA. n=10

SUMMARY:
The important role of mechanical joint stress for the insert and progress of osteoarthritis (OA) is supported by recent studies. The degeneration of joint cartilage is caused either by unphysiological load of a healthy joint or physiological load of a damaged joint. The exact mechanisms leading from increased weight bearing and overuse to cartilage degeneration are mostly unknown.

The hypothesis of the study is that parameters of oxidative stress in the joint synovial space reflect damages possibly leading to OA. These parameters correlate with parameters of oxidative stress in the peripheral blood. Aim of the study is the identification of such non- invasive obtainable biomarkers which represent the degenerative and regenerative changes in joint.

DETAILED DESCRIPTION:
Patients with clinically manifest OA typically consult the physician at time of irreversible cartilage destruction. This is due to the long time clinically silent progress of the disease. A biomarker screening profile for joint damage is a valuable tool for the detection of over use and joint damaging conditions especially in competitive sports. This would provide a method for OA risk assessment for the patient before clinical symptoms occur. For this the first step is the identification of biological substances reflecting pathologic changes in the joint.

Since preterm chondrocyte senescence, apoptosis and ageing related changes are key factors in OA pathophysiology and each of these factors is closely related to oxidative dysbalance the measurement of these factors and correlation with the amount of joint damage is promising.

ELIGIBILITY:
Inclusion Criteria:

* Planned knee joint arthroscopy
* No history of trauma

Exclusion Criteria:

* Neoplasia
* Rheumatoid arthritis
* Intake of Steroids, cytostatic drugs,immunosuppression
* Pregnancy or lactation
* Addiction
* Participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University clinic, patients, residents of Düsseldorf, Germany and surrounding cities
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Department, Heinrich-Heine University Medical School, Düsseldorf, North Rhine-Westphalia, Germany